CLINICAL TRIAL: NCT02203851
Title: An Open Label Extension Trial Assessing the Safety and Efficacy of BI 655066/ ABBV-066/Risankizumab Administered Subcutaneously in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Extension Trial Assessing the Safety and Efficacy of BI 655066/ABBV-066/Risankizumab in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-009; 2014-001687-36 (EudraCT Number); 1311.13 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Psoriasis
Keywords: BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risankizumab 90 mg (Experimental): Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had achieved ≥90% improvement in Psoriasis Area and Severity Index (PASI90) Score at Week 12 continued to receive open-label (OL) risankizumab 90 mg by SC injection at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
  Interventions: Drug: Risankizumab
- Risankizumab 180 mg (Experimental): Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had achieved <90% improvement in Psoriasis Area and Severity Index (PASI90) Score at Week 12 switched to open-label (OL) risankizumab 180 mg by SC injection at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab administered by subcutaneous (SC) injection
  Other Names: BI 655066; ABBV-066; SKYRIZI

SUMMARY:
The primary objective of Study M16-009 was to investigate the safety of risankizumab in participants with moderate to severe chronic plaque psoriasis who were receiving long-term treatment. Additional study objectives were to further investigate the long-term efficacy, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of risankizumab.

DETAILED DESCRIPTION:
Participants who had successfully completed Study 1311.2 (NCT02054481; the lead-in study) and met the eligibility criteria for Study M16-009 (extension study) had the option to enter the extension study. Participants were allowed to have the End of Study Visit in the lead in study combined with the Week 0 Visit for the extension study. At the Week 12 visit, participants were assigned to treatment based on 90% improvement in Psoriasis Area and Severity Index (PASI90) Score: participants with ≥PASI90 Score at Week 12 continued to receive risankizumab 90 mg by subcutaneous (SC) injection; participants with <PASI90 Score at Week 12 switched to risankizumab 180 mg by SC injection.

Efficacy results are summarized by the 4 treatment groups from the lead-in study, which included the following: Participants who received risankizumab 18 mg in the lead-in study and risankizumab in the extension study (Risankizumab 18 mg/Risankizumab); participants who received risankizumab 90 mg in the lead-in study and risankizumab in the extension study (Risankizumab 90 mg/Risankizumab); participants who received risankizumab 180 mg in the lead-in study and risankizumab in the extension study (Risankizumab 180 mg/Risankizumab); and participants who received ustekinumab (Stelara) 45 or 90 mg in the lead-in study and risankizumab in the extension study (Ustekinumab/Risankizumab).

ELIGIBILITY:
Inclusion criteria:

* Participants with moderate to severe chronic plaque psoriasis, who have successfully completed Study 1311.2 (NCT02054481; the lead-in study). Successful completion of the lead-in study is defined as either of the following:

  1. Completion of the entire follow up period, thus reaching End-of-study (EOS) visit.
  2. Loss of response, defined as decrease in response to achieving < 50% improvement in Psoriasis Area and Severity Index Score (PASI50) at any time from Week 24.
* Participant must give informed consent and sign an approved consent form prior to any study procedures in accordance with Good Clinical Practice (GCP) and local legislation
* Applicable only for female participants:
* Negative urine pregnancy dip stick test at the roll-over visit, and if available at roll-over visit, negative Serum ß-Human Chorionic Gonadotropin (ß-HCG) test.

In addition:

Women of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopausal), that, if sexually active agree to use one of the appropriate medically accepted methods of birth control in addition to the consistent and correct use of a condom from date of the roll-over visit until 12 weeks after last treatment in this study. Medically accepted methods of contraception are: ethinyl estradiol containing contraceptives, diaphragm with spermicide substance, and intra-uterine-device.

OR

Female participants which have vasectomized sexual partner(s) (vasectomy at least 1 year prior to enrollment).

OR

Surgically sterilized female participants with documentation of prior hysterectomy, tubal ligation or complete bilateral oophorectomy.

OR

Postmenopausal women with postmenopausal is defined as permanent cessation ≥ 1 year of previously occurring menses.

Exclusion criteria:

* Participants who experienced any drug related serious adverse event (SAE) in the lead-in study
* Participants who have developed guttate, erythrodermic or pustular psoriasis or drug-induced psoriasis (as diagnosed by the investigator), during the lead-in study.
* Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and electrocardiography [ECG]), that in the opinion of the investigator, would compromise the safety of the participant or the quality of the data.
* Known clinically important acute or chronic infections including hepatitis, human immunodeficiency virus (HIV). In regards to tuberculosis (TB), the following applies:
* Signs or symptoms suggestive of current active or latent TB upon medical history, physical examination and/or a chest radiograph (both posterior-anterior and lateral views, taken within 3 months prior to the first administration of study drug and read by a qualified radiologist).
* History of latent or active TB prior to screening, except for participants with documented completion of an adequate treatment regimen, at least 6 months prior to the first administration of study agent.
* Positive QuantiFERON-TB Gold In-Tube test (IGRA) within 2 months prior to the roll-over visit (if available), in which active TB has not been ruled out. This does not apply to participants with history of latent TB with documented completion of an adequate treatment regimen, at least 6 months prior to the first administration of study agent.
* Participants who have developed malignancy, or suspicion of active malignant disease during the lead-in study (except treated cutaneous squamous cell or basal cell carcinoma or carcinoma in situ of the cervix that have been adequately treated).
* Intake of restricted medications or other drugs considered likely to interfere with the safe conduct of this study, as assessed by the investigator.
* Alcohol or drug abuse within 3 months prior to the roll-over visit that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures in the opinion of the investigator.
* Any clinically significant laboratory abnormalities based on the last available laboratory results received during the lead-in study (according to the investigator's medical assessment).
* Pre-menopausal woman who is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Papp KA, de Vente S, Zeng J, Flack M, Padilla B, Tyring SK. Long-Term Safety and Efficacy of Risankizumab in Patients with Moderate-to-Severe Chronic Plaque Psoriasis: Results from a Phase 2 Open-Label Extension Trial. Dermatol Ther (Heidelb). 2021 Apr;11(2):487-497. doi: 10.1007/s13555-021-00490-3. Epub 2021 Jan 29. PMID 33512666
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analyses were performed using the intent-to-treat (ITT) population defined as all participants who received at least 1 dose of study drug. As predefined, the demographics, disposition and safety results were summarized for ITT population. Efficacy results were summarized by the 4 treatment groups from the lead-in study (Study 1311.2; NCT02054481).
Pre-assignment Details: Participants completing lead-in study and met eligibility for this study were enrolled; demographic/disposition were not collected by dose level. Some participants in extension study had dose escalation due to lack of efficacy, predefined selected safety analysis were broken down by groups: participants remaining at 90mg and those receiving 180mg.
Groups:
- Risankizumab 90 mg or 180 mg: Participants received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
Period: Overall Study
Arm/Group | Risankizumab 90 mg or 180 mg
Started | 110
Completed | 99
Not Completed | 11
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 6
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: All participants that received at least one dose of study drug in the extension study who either remained at 90 mg throughout the study or who received 180 mg were summarized.
Arm/Group | Risankizumab 90 mg or 180 mg
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 2
  White | 101
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event with an onset after the first dose of risankizumab in this study. See the Adverse Event section for details.
Time Frame: From first dose of study drug in either the lead-in or extension study until 12 weeks after the last dose of study drug (approximately 4 years from the first dose in either the lead-in or extension study)
Population: Safety population, which is the same as the Intent to Treat (ITT) population for this study (defined as all participants who received at least one dose of study drug in the study), summarized by the group the participants who remained at 90 mg throughout the study and the participants who received 180 mg
Measure: Number; unit: participants
Groups:
- Risankizumab 90 mg: Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had ≥ PASI 90 at week 12 continued to receive risankizumab 90 mg at Week 12 and every 12 weeks for 4 years.
- Risankizumab 180 mg: Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had < PASI 90 at week 12 switched to risankizumab 180 mg at Week 12 and every 12 weeks for 4 years.
Arm/Group | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 87 | 23
participants | 67 | 18

2. Primary Outcome: Number of Participants With Drug-related TEAEs
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Safety Population summarized by the group the participants who remained at 90 mg throughout the study and the participants who received 180 mg
Measure: Number; unit: participants
Arm/Group | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 87 | 23
participants | 12 | 3

3. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Risankizumab 90 mg | Risankizumab 180 mg
Number analyzed (Participants) | 87 | 23
participants | 12 | 2

4. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI90) Score at Week 48 in the Extended Dosing Period
Description: Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. Baseline PASI for this study is defined as the baseline PASI in the lead-in study. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 48
Population: ITT population: defined as all participants who received at least one dose of study drug in the study and summarized by the 4 treatment groups from the lead-in study (Study 1311.2; NCT02054481).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Risankizumab 18 mg/Risankizumab: Participants who received risankizumab 18 mg in the lead-in study received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection in this study at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
- Risankizumab 90 mg/Risankizumab: Participants who received risankizumab 90 mg in the lead-in study received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection in this study at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
- Risankizumab 180 mg/Risankizumab: Participants who received risankizumab 180 mg in the lead-in study received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection in this study at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
- Ustekinumab/Risankizumab: Participants who received ustekinumab 45 mg or 90 mg in the lead-in study received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection in this study at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 72.7 [54.1 to 91.3] | 77.8 [62.1 to 93.5] | 71.9 [56.3 to 87.5] | 74.1 [57.5 to 90.6]

5. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of Clear or Almost Clear at Week 48 of Extended Dosing Period
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. Baseline is defined as the last non-missing value on or before the date of the first dose of study drug in the lead-in study.
Time Frame: Week 48
Population: ITT Population summarized by the 4 treatment groups from the lead-in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 63.6 [43.5 to 83.7] | 70.4 [53.1 to 87.6] | 68.8 [52.7 to 84.8] | 66.7 [48.9 to 84.4]

6. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in PASI (PASI50) Score at Week 48 in the Extended Dosing Period
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI50 is defined as at least a 50% reduction in PASI score compared with the Baseline PASI score. Baseline PASI for this study is defined as the baseline PASI in the lead-in study. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 48
Population: ITT population summarized by the 4 treatment groups from the lead-in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Risankizumab 18 mg/Risankizumab: Participants who received risankizumab 18 mg in the lead-in study received open-label (OL) risankizumab 90 mg or 180 mg by subcutaneous (SC) injection in this study at Week 12 and every 12 weeksfor approximately 4 years from the first dose in either the lead-in or extension study.
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 95.5 [86.8 to 100.0] | 96.3 [89.2 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI (PASI75) Score at Week 48 in the Extended Dosing Period
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. Baseline PASI for this study is defined as the baseline PASI in the lead-in study. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 48
Population: ITT population summarized by the 4 treatment groups from the lead-in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 86.4 [72.0 to 100.0] | 92.6 [82.7 to 100.0] | 90.6 [80.5 to 100.0] | 96.3 [89.2 to 100.0]

8. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI (PASI100) Score at Week 48 in the Extended Dosing Period
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. Baseline PASI for this study is defined as the baseline PASI in the lead-in study. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 48
Population: ITT population summarized by the 4 treatment groups from the lead-in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 54.5 [33.7 to 75.4] | 55.6 [36.8 to 74.3] | 50.0 [32.7 to 67.3] | 55.6 [36.8 to 74.3]

9. Secondary Outcome: Percentage of Participants Achieving sPGA of Clear at Week 48 of Extended Dosing Period
Description: as for outcome 5
Time Frame: Week 48
Population: ITT Population summarized by the 4 treatment groups from the lead-in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab 18 mg/Risankizumab | Risankizumab 90 mg/Risankizumab | Risankizumab 180 mg/Risankizumab | Ustekinumab/Risankizumab
Number analyzed (Participants) | 22 | 27 | 32 | 27
percentage of participants | 54.5 [33.7 to 75.4] | 63.0 [44.7 to 81.2] | 56.3 [39.1 to 73.4] | 55.6 [36.8 to 74.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug in either the lead-in or extension study with an onset date within 105 days after the last dose of study drug or approximately 4 years from the first dose in either the lead-in or extension study.
Groups:
- Risankizumab 90 mg: Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had ≥ PASI 90 at week 12 continued to receive risankizumab 90 mg at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
- Risankizumab 180 mg: Participants entered the study receiving risankizumab 90 mg by subcutaneous (SC) injection and had < PASI 90 at week 12 switched to risankizumab 180 mg at Week 12 and every 12 weeks for approximately 4 years from the first dose in either the lead-in or extension study.
Arm/Group | Risankizumab 90 mg | Risankizumab 180 mg
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/23
Serious Adverse Events (participants affected / at risk) | 12/87 | 2/23
Other Adverse Events (participants affected / at risk) | 46/87 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 90 mg (N=87) | Risankizumab 180 mg (N=23)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (3) | 0 (0)
Ulnar neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 90 mg (N=87) | Risankizumab 180 mg (N=23)
Bronchitis (Infections and infestations) | 5 (6) | 2 (2)
Influenza (Infections and infestations) | 7 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 16 (33) | 3 (8)
Sinusitis (Infections and infestations) | 3 (5) | 3 (3)
Tooth abscess (Infections and infestations) | 6 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (16) | 4 (5)
Urinary tract infection (Infections and infestations) | 8 (9) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02203851/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02203851/SAP_001.pdf